CLINICAL TRIAL: NCT06057415
Title: Improving Gastrointestinal Function In High-Risk Newborns By Stimulation Of The Enteric Nervous System
Acronym: NeoHemoHapt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114536
Record Dates: First submitted 2023-06-21; First posted 2023-09-28 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-06

CONDITIONS: Feeding and Eating Disorders
Keywords: preterm infants; high-risk newborns; congenital diaphragmatic hernia; autonomous nervous system; tactile stimulation
MeSH Terms: conditions — Feeding and Eating Disorders; Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Intervention Model Description: The randomization will occur web-based, and will be protected from selection bias by using concealed, stratified and blocked randomization.
  The group of preterm infants will randomly be assigned to 2 treatment groups according to 6 strata.
  * Gestational age 24+0 - 26+0 weeks + Appropriate for gestational age (AGA)
  * Gestational age 24+0 - 26+0 weeks + Small for gestational age (SGA)
  * Gestational age 26+1 - 28+0 weeks + AGA
  * Gestational age 26+1 - 28+0 weeks + SGA
  * Gestational age 28+1 - 29+6 weeks + AGA
  * Gestational age 28+1 - 29+6 weeks + SGA
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Will receive standard of care according to the institutional protocol and principles of developmental care which currently belongs to (inter-) national guidelines and is regarded as safe.
- Standard care supplemented with HAPTOS intervention (Experimental): Will receive standard of care according to the principles of developmental care which currently belongs to (inter-) national guidelines plus HAPTOS intervention which includes: tactile/ kinaesthetic massage of the trunk and extremities twice daily and stimulation of oral function by providing perioral stimulation up to 4 times a day. Interventions will be continued until clinical improvement.
  Interventions: Procedure: HAPTOS (Handling Adapted to Postnatal age with Tactile-kinaesthetic and Oral sensorimotor Stimulation

INTERVENTIONS:
Procedure: HAPTOS (Handling Adapted to Postnatal age with Tactile-kinaesthetic and Oral sensorimotor Stimulation — Tactile-kinaesthetic and Oral sensorimotor Stimulation
  Arms: Standard care supplemented with HAPTOS intervention

SUMMARY:
The goal of this therapeutical intervention trial is to investigate whether tactile-kinesthaetic and oral sensorimotor stimulation can improve gastrointestional function in preterm infants born before gestational age of 30 weeks and newborns with congenital diaphragmatic hernia. The main question it aims to answer is:

• To determine whether HAPTOS- intervention (Handling Adapted to Postnatal age with Tactile-kinaesthetic and Oral sensorimotor Stimulation) in the particpants results in earlier attainment (postnatal days) of full enteral feeding and/or full oral feeding (post menstrual age) compared to standard care. Researchers will compare an intervention group receiving standard of care plus HAPTOS intervention to a group of patients receiving only current standard of care.

DETAILED DESCRIPTION:
Infants born preterm or with congenital diaphragmatic hernia (CDH) are at risk for several long-term unfavourable outcomes that can be related to feeding difficulties from birth onwards. Adverse nutritional outcomes in both patient groups mainly originate from mechanical dysfunction, based on dysmotility. Mechanical function includes suck-swallow coordination, gastrointestinal sphincter tone, gastric emptying and intestinal motility and is regulated by the complex interplay of the autonomic (ANS) and enteric (ENS) nervous system with modulation by the central nervous system (CNS). The intra-uterine environment provides the fetus with developmentally timed sensory exposures through 'touch' that are necessary for development of sensory control and autonomous coordination of bodily functions. Preterm infants miss out this normal maturation, while newborns with CDH may exhibit a delayed maturation probably as a result of the deviant anatomical situation and the severe illness during the direct postnatal period. In the postnatal situation both patient groups may be confronted with either 'negative' sensory stimulation through exposures such as procedural touch/handling, pain or otherwise a reduction in sensory exposures through avoidance of positive touch in relation to supposed clinical instability. All together this may affect normal development and may lead to sensory deprivation and delayed maturation of the nervous regulation and cerebral maturation. Tactile-kinaesthetic and oral sensorimotor stimulation using positive gentle touch have been shown to positively affect cardiorespiratory stability, weight gain, gastro-intestinal performance, and length of stay in hospital for preterm infants. However, these strategies have not been evaluated in high-risk infants. The current study aims at evaluating an intervention programme that provides positive stimuli through touch adapted to the stage of development of the infant with regard to timing, duration and intensity that supports the maturational development of gastrointestinal functionality. (Handling Adapted to Postnatal age with Tactile-kinaesthetic and Oral sensorimotor Stimulation; HAPTOS intervention). We hypothesize that the HAPTOS intervention will improve the postnatal maturation of the autonomous and enteral nervous system and cause improvements in gastrointestinal motility, enteral and oral feeding and cardiorespiratory stability.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm birth at gestational age < 30 weeks or
2. Diagnosis of Congenital Diaphragmatic Hernia
3. Born at Amalia Children's Hospital or admitted 1rst day of life
4. Written informed consent of both parents or representatives

Exclusion Criteria:

1. Preterm infant born at gestational age ≥ 30 weeks
2. Perinatal Asphyxia; (Apgar score at 5' < 5 and first pH ≤ 7,0)
3. Major congenital anomalies or birth defects other than congenital diaphragmatic hernia;
4. Metabolic disease that necessitates a special diet other than human milk or formula feeding and or has a prognosis of impaired neurological development
5. Parental refusal of participation

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of days to achieve full enteral feeding | 60 days
  measuring the time from birth until enteral intake reaches 150ml/kg/d
Postmenstrual age at achievement of full oral feeding | 52 weeks
  Number of postmenstrual weeks until gastrointestinal tube is taken out

SECONDARY OUTCOMES:
First meconium passage | 14 days
  Postnatal day at first meconium
Duration of meconium passage | 14 days
  Number of days until normal defecation
Use of laxatives | 60 days
  Number of laxatives given
Gastrointestinal Motility | 100 days
  Volume of gastric residuals per week
Vomiting | duration of hospitalization up to 15 months
  Number of incidences of vomiting in combination with aspiration
Periodic breathing | duration of hospitalization up to 15 months
  Number of desaturations < 80% and/or bradycardia < 80/min that require intervention per week
Feeding difficulties | 24 months
  Number of infants with impaired oral motor skills
Maturation of heart rate variability | duration of intensive care stay up to 60 days
  Number of infants with delayed regulation of the para- and sympathicus tonus measured continuously through monitordata collection
Growth at postmenstrual age | at 40 weeks, 3, 6, 12, 18 and 24 weeks
  Gain in weight, length, and head circumference including percentiles
Morbidity | 100 days
  Number of infants with necrotizing enterocolitis, spsis, chronic lung disease, retinopathy of prematurity, intra-ventricular hemorrhage
Duration hospital stay | 100 days
  Postnatal age at time of discharge home
Neurocognitive development | at 24 months
  Measuring cognitive and motor development using Bayley Scores of Infant Development (BSID III)
Parent participation in care | duration of hospitalization up to 100 days
  Measuring number of parents who participate and frequency of activity

CONTACTS AND LOCATIONS:
Overall Officials: Viola Christmann, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands